CLINICAL TRIAL: NCT04965272
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Fixed-Dose, Phase 2 Study Evaluating the Safety and Efficacy of Cariprazine as an Adjunctive Therapy to Antidepressant Therapies (ADTs), in the Treatment of Subjects With Generalized Anxiety Disorder (GAD) Who Have Had an Inadequate Response to ADT Alone
Brief Title: A Study To Assess Adverse Events and Change in Disease Activity With Oral Cariprazine When Added to Antidepressant Therapies (ADTs) Compared to Placebo in Adult Participants With Generalized Anxiety Disorder (GAD) Who Have Had an Inadequate Response to ADTs Alone
Acronym: CAR aGAD Ph 2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-209
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder (GAD); Cariprazine; Vraylar; Depression; Antidepressant therapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Depression | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cariprazine 0.75 mg/day + Antidepressant Therapy (Experimental): Antidepressant (paroxetine, escitalopram, venlafaxine XR, or duloxetine) + cariprazine 0.75 mg/day oral, once daily for 6 weeks
  Interventions: Drug: Cariprazine 0.75 mg/day
- Cariprazine 1.5 mg/day + Antidepressant Therapy (Experimental): Antidepressant (paroxetine, escitalopram, venlafaxine XR, or duloxetine) + cariprazine 1.5 mg/day oral, once daily for 6 weeks
  Interventions: Drug: Cariprazine 1.5 mg/day
- Cariprazine 3.0 mg/day + Antidepressant Therapy (Experimental): Antidepressant (paroxetine, escitalopram, venlafaxine XR, or duloxetine) + cariprazine 1.5 mg/day oral for 2 weeks followed by cariprazine 3.0 mg/day oral, once daily for 4 weeks.
  Interventions: Drug: Cariprazine 3.0 mg/day
- Placebo + Antidepressant Therapy (Placebo Comparator): Antidepressant (paroxetine, escitalopram, venlafaxine XR, or duloxetine) + oral placebo, once daily for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cariprazine 0.75 mg/day — Oral Capsule
  Other Names: Vraylar
  Arms: Cariprazine 0.75 mg/day + Antidepressant Therapy
Drug: Cariprazine 1.5 mg/day — Oral Capsule
  Other Names: Vraylar
  Arms: Cariprazine 1.5 mg/day + Antidepressant Therapy
Drug: Cariprazine 3.0 mg/day — Oral Capsule
  Other Names: Vraylar
  Arms: Cariprazine 3.0 mg/day + Antidepressant Therapy
Other: Placebo — Oral Capsule
  Arms: Placebo + Antidepressant Therapy

SUMMARY:
Generalized anxiety disorder (GAD) is usually treated with antidepressant therapy (ADT); however, sometimes ADTs alone are not enough to adequately treat GAD. The purpose of this study is to assess adverse events and the change in disease activity with cariprazine when added to ADTs compared with placebo in adult participants with GAD who have had an inadequate response to 1 or more prior ADTs alone.

Cariprazine is an approved drug being developed for the treatment of GAD. The participants are placed into 1 of 4 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 4 chance that participants will be assigned to placebo. Around 1072 participants age 18-65 with GAD and an inadequate response to ADT alone will be enrolled in the study in the United States.

After a 2-week screening period, participants will receive daily oral capsules of cariprazine of varying doses or placebo for 6 weeks, followed by a 4-week safety follow-up period for a total study duration of 10 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants with generalized anxiety disorder (GAD).
* Taking one of the FDA-approved antidepressant therapies (ADTs) for the treatment of GAD (i.e., escitalopram, paroxetine, duloxetine, and venlafaxine XR).
* Continuing to exhibit anxiety symptoms (Hamilton Anxiety Scale [HAM-A] total score >= 22) at Visit 1 (Screening) and Visit 2 (Baseline, Week 0) despite being on an adequate dose and duration (at least 6 weeks of continuous use, with a minimum of 3 of 6 weeks above the minimum labeled dose for GAD).
* Documentation of inadequate response to at least 1 ADT must be confirmed on the GAD-Antidepressant Treatment Response Questionnaire (GAD-ATRQ).
* Must have a minimum score of 22 on the rater-administrated HAM-A and a minimum score of 4 on the rater-administered Clinical Global Impression of Severity Scale (CGI-S), at both Visit 1 (Screening) and Visit 2 (Baseline, Week 0).
* A score of less than 12 on the rater-administered Hamilton Depression Rating Scale-17-item (HAMD-17) at Visit 1 (Screening) and Visit 2 (Baseline, Week 0).
* Laboratory values must meet the criteria specified in the protocol within the screening period prior to the first dose of study drug.

Exclusion Criteria:

* Psychiatric comorbidities, risk of suicide, self-injury, and/or harm to others; any current Diagnostic and Statistical Manual of Mental Disorders - 5th edition (DSM-5) psychiatric diagnosis other than generalized anxiety disorder (GAD) (other than specific phobias) or history of alcohol or any other substance-related disorders within the 6 months before Visit 1 (Screening).
* Pregnancy, current breastfeeding status, plans to become pregnant or to donate eggs during the study or for approximately 30 days after the last dose of investigational product (female participants).
* History of an allergic reaction, hypersensitivity, or intolerance to constituents of cariprazine (and its excipients) and/or other products of the same class or to any of the protocol-approved rescue medications.
* Any clinically relevant or significant electrocardiogram (ECG) abnormalities, including ECG with QT interval corrected for heart rate (QTc) using Fridericia's formula (QTcF) >450 msec (males) or >470 msec (females).
* History of seizure disorder, with the exception of febrile seizure, stroke, significant head injury, tumor of the central nervous system, or any other condition that predisposes to seizure.
* Specific medical conditions precluding study drug use and/or study participation, such as history of neuroleptic malignant syndrome; cataracts or retinal detachment; allergic reactions/hypersensitivity to cariprazine and/or protocol-approved rescue medications; pregnancy per above; cardiovascular disease; seizure history; and any other disease that is clinically unstable or would make the participant an unsuitable candidate to participate in the study, based on the investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-18 (Estimated); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score | Week 6
  The HAM-A is a 14-item, clinician-reported measure used to quantify and categorize the participant's anxiety over the past week. Items are rated on a 5-point Likert rating scale. The HAM-A total score ranges from 0 to 56, with higher scores indicating greater anxiety severity.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Global Impression of Severity Scale (CGI-S) | Week 6
  The CGI-S is a single, clinician-reported item that measures the clinician's impression of a subject's current anxiety severity considering their total clinical experience with the patient population. The measure uses a 5-point Likert rating scale, with higher scores indicating greater anxiety severity.
Percentage of Participants in Remission | Week 6
  Remission is defined as HAM-A total score <=7, Clinical Global Impression of Improvement Scale (CGI-I) = 1, and Sheehan Disability Scale: Anxiety (SDS: Anxiety) total score <= 5
Percentage of Participants with HAM-A Response | Week 6
  HAM-A response is defined as >= 50% reduction from baseline in HAM-A total score
Percentage of Participants with CGI-I Responder Status of "Much Better" or "Very Much Better" | Week 6
  The CGI-I is a single, clinician reported item that measures the clinician's impression of how much a participant's anxiety has changed since starting the study medication compared to the participant's condition at baseline. The measure uses a 7-point Likert rating scale with responses ranging from "very much better" (1) to "very much worse" (7).
Percentage of Participants with Patient Global Impression of Change Scale (PGI-C) Responder Status of "Much Better" or "Very Much Better" | Week 6
  The PGI-C is a single, patient-reported item that assesses the participant's perceived overall change in their anxiety since they started taking the study medication. The measure uses a 7-point Likert rating scale with responses ranging from "very much better" (1) to "very much worse" (7).
Change from Baseline in Patient Global Impression of Severity Scale (PGI-S) | Week 6
  The PGI-S is a single, patient-reported item that assesses the participant's perceived level of anxiety over the past 7 days. The measure uses a 5-point Likert rating scale with responses ranging from "none" (1) to "very severe" (5), with higher scores indicating greater anxiety severity.
Change from Baseline in SDS: Anxiety Total Score | Week 6
  The SDS: Anxiety is a 5-item, patient-reported measure used to assess functional impairment in the domains of work/school, social life, and family life on a 10-point numeric rating scale with verbal anchors. The 3 items assessing work/school, social life, and home life or family responsibilities impairment are summed into a single dimensional measure of global functional impairment, with scores ranging from 0 (unimpaired) to 30 (highly impaired). Higher scores indicate greater impairment.
Change from Baseline in Hamilton Depression Rating Scale-17 item, via Structured Interview Guide for the Hamilton Depression Scale (HAMD-17) Total Score | Week 6
  The HAMD-17 is a 17-item, clinician-reported measure used to quantify and categorize the participant's depression over the past week. The HAMD-17 total score ranges from 0 to 52 with higher scores indicating greater depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (36):
- United States (36):
  - Preferred Research Partners /ID# 232286, Little Rock, Arkansas
  - Axiom Research /ID# 230728, Colton, California
  - ATP Clinical Research, Inc /ID# 230445, Costa Mesa, California
  - ProScience Research Group /ID# 231520, Culver City, California
  - WR-PRI, LLC - Encino /ID# 230434, Encino, California
  - Synergy San Diego /ID# 231006, Lemon Grove, California
  - Pharmacology Research Institute - Wake LLC /ID# 230722, Los Alamitos, California
  - Pharmacology Research Inst /ID# 230869, Newport Beach, California
  - Anderson Clinical Research /ID# 230440, Redlands, California
  - California Neuroscience Research Medical Group, Inc. /ID# 230453, Sherman Oaks, California
  - Viking Clinical Research /ID# 230379, Temecula, California
  - Pacific Clinical Research Management Group /ID# 229725, Upland, California
  - Galiz Research - Palmetto Medical Plaza /ID# 230446, Hialeah, Florida
  - Great Lakes Clinical Trials /ID# 231296, Chicago, Illinois
  - Baber Research Group /ID# 230447, Naperville, Illinois
  - Boston Clinical Trials /ID# 231003, Boston, Massachusetts
  - ActivMed Practices and Research, LLC. /ID# 230441, Methuen, Massachusetts
  - Alivation Research /ID# 230449, Lincoln, Nebraska
  - Center for Emotional Fitness /ID# 230450, Cherry Hill, New Jersey
  - Hassman Research Institute Marlton /ID# 233252, Marlton, New Jersey
  - Integrative Clinical Trials /ID# 230955, Brooklyn, New York
  - SPRI Clinical Trails /ID# 230957, Brooklyn, New York
  - Fieve Clinical Research, Inc. /ID# 230452, New York, New York
  - Clinilabs, Inc. /ID# 230958, New York, New York
  - Manhattan Behavioral Medicine PLLC /ID# 229713, New York, New York
  - Carolina Institute for Clinical Research - Fayetteville /ID# 230961, Fayetteville, North Carolina
  - Ohio State Harding Hospital /ID# 231302, Columbus, Ohio
  - CincyScience /ID# 229719, West Chester, Ohio
  - Sooner Clinical Research /ID# 229731, Oklahoma City, Oklahoma
  - Research Strategies of Memphis /ID# 230443, Memphis, Tennessee
  - Clinical Neuroscience Solutions - Memphis /ID# 230734, Memphis, Tennessee
  - Austin Clinical Trial Partners /ID# 229727, Austin, Texas
  - FutureSearch Trials of Dallas, LP /ID# 230535, Dallas, Texas
  - Earle Research /ID# 230969, Houston, Texas
  - Grayline Research Center /ID# 230455, Wichita Falls, Texas
  - Woodstock Research Center /ID# 231005, Woodstock, Vermont

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com